CLINICAL TRIAL: NCT03092089
Title: Sonothrombolysis in Patients With an ST-segment Elevation Myocardial Infarction. A Prospective Single-arm Study.
Brief Title: Sonothrombolysis in Patients With STEMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harald Becher (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Harald Becher, Professor of Medicine, University of Alberta
Organization: University of Alberta (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST2017-Pro00067953; Pro00067953 (Other: Health Ethics Research Board)
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: Sonothrombolysis, STEMI, PPCI, Microbubbles
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: This clinical study is a prospective single-center, single-arm investigation of sonothrombolysis in adult patients presenting with high-risk STEMI within 6 hrs of the onset of clinical symptoms and receiving reperfusion therapy with PCI. All patients will receive standard therapy. Patients will immediately receive an iv infusion of commercially available ultrasound contrast agent (Definity) and myocardial contrast echocardiography will be performed to document the size of the perfusion defect. Loops of 15 cardiac cycles will be recorded using low mechanical index (MI) ultrasound. These recordings will also be used to assess regional wall motion as well as LV volumes and ejection fraction. Immediately after the diagnostic ultrasound, the therapeutic ultrasound will start using the same transducer by applying multiple high MI ultrasound impulses. These pulses will be applied to the apical windows that contained the risk area. The intervals between HMI impulses will vary from 5 to 15 s.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adult patients with high risk STEMI (Experimental): Adult patients presenting with high-risk STEMI will receive sonothrombolysis with Definity in addition to standard of care (reperfusion therapy with PPCI)
  Interventions: Drug: Definity, (Lipid Microspheres) Intravenous Suspension; Device: Myocardial Contrast Echocardiography; Procedure: Repurfusion therapy with PPCI

INTERVENTIONS:
Drug: Definity, (Lipid Microspheres) Intravenous Suspension — Sonothrombolysis (High Impulse therapeutic ultrasound with infusion of ultrasound contrast agent Definity) will be applied before and after standard of care reperfusion therapy with PPCI
Device: Myocardial Contrast Echocardiography — Myocardial contrast echocardiography will be applied before standard of care reperfusion therapy as well as prior to discharge and at 3 month follow up
Procedure: Repurfusion therapy with PPCI — Patients will receive reperfusion therapy with PPCI as standard of care

SUMMARY:
This study evaluates what effect sonothrombolysis may have on spontaneous reperfusion, microvascular obstruction, left ventricular function and infarct size in patients presenting with their first ST-segment Elevation Myocardial Infarction.

DETAILED DESCRIPTION:
This is a prospective, single center, single-arm study that examines pre-procedural sonothrombolysis as an adjuvant to contemporary therapy in patients with ST-segment elevation myocardial infarction receiving PPCI.This study is to examine what effect adding emergent diagnostic ultrasound (DUS) guided high mechanical index (HMI) impulses (sonothrombolysis), applied both before and after primary percutaneous coronary intervention (PPCI) during an intravenous commercially available microbubble infusion (Definity), have on spontaneous reperfusion (i.e. pre PCI coronary artery patency rates), microvascular obstruction, left ventricular function and infarct size in patients presenting with their first ST-segment Elevation Myocardial Infarction.

Patients will immediately receive an intravenous infusion of commercially available ultrasound contrast agent (Definity). After starting the infusion, myocardial contrast echocardiography will be performed. 4-, 2- and 3-chamber views will be recorded to document the size of the perfusion defect. Loops of 15 cardiac cycles will be recorded using low mechanical index (MI) ultrasound with a 'flash' delivered after the second cardiac cycle of the loop. The flash is a short impulse of HMI ultrasound which is transmitted to destroy the ultrasound contrast in the myocardium and then to assess the replenishment of myocardial contrast. These recordings will also be used to assess regional wall motion as well as the LV volumes and ejection fraction. Immediately after the diagnostic ultrasound, the therapeutic ultrasound will start using the same transducer by applying multiple HMI ultrasound impulses. The HMI are the same as those which are used for assessment of myocardial perfusion in diagnostic ultrasound. These pulses will be applied in the apical 4-, 2-, and 3-chamber views to the apical windows that contained the risk area. The intervals between HMI impulses will vary from 5 to 15 s depending on the time required for myocardial contrast replenishment. Diagnostic echocardiography will also be scheduled prior to discharge (Day2) and 90 days post procedure.

If this study is successful, a larger study will be designed in order to collect the evidence for using contrast ultrasound for treatment of myocardial infarction in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with STEMI within 6 hours of symptom onset and:

1. Are expected to receive reperfusion therapy with primary PCI
2. Have a high-risk STEMI ECG defined as:

   * ≥2mm ST-segment elevation in 2 anterior or lateral leads; or
   * ≥2 mm ST-segment elevation in 2 inferior leads coupled with ST segment depression in 2 contiguous anterior leads for a total ST-segment deviation of ≥4mm
3. Age ≥30 years.
4. Adequate apical and/or parasternal images by echocardiography

Exclusion Criteria:

1. Isolated inferior STEMI without anterior ST-segment depression
2. Previous coronary bypass surgery
3. Cardiogenic shock
4. Known or suspected hypersensitivity to ultrasound contrast agent used for the study
5. Life expectancy of less than two months or terminally ill.
6. Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors, anticoagulants, or aspirin
7. Known large right to left intracardiac shunts.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Becher, Principal Investigator — University of Alberta
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slikkerveer J, Kleijn SA, Appelman Y, Porter TR, Veen G, van Rossum AC, Kamp O. Ultrasound enhanced prehospital thrombolysis using microbubbles infusion in patients with acute ST elevation myocardial infarction: pilot of the Sonolysis study. Ultrasound Med Biol. 2012 Feb;38(2):247-52. doi: 10.1016/j.ultrasmedbio.2011.11.001. Epub 2011 Dec 16. PMID 22178160
- [Background] Xie F, Lof J, Everbach C, He A, Bennett RM, Matsunaga T, Johanning J, Porter TR. Treatment of acute intravascular thrombi with diagnostic ultrasound and intravenous microbubbles. JACC Cardiovasc Imaging. 2009 Apr;2(4):511-8. doi: 10.1016/j.jcmg.2009.02.002. PMID 19580735
- [Background] Roos ST, Juffermans LJ, van Royen N, van Rossum AC, Xie F, Appelman Y, Porter TR, Kamp O. Unexpected High Incidence of Coronary Vasoconstriction in the Reduction of Microvascular Injury Using Sonolysis (ROMIUS) Trial. Ultrasound Med Biol. 2016 Aug;42(8):1919-28. doi: 10.1016/j.ultrasmedbio.2016.03.032. Epub 2016 May 6. PMID 27160847
- [Background] Mathias W Jr, Tsutsui JM, Tavares BG, Xie F, Aguiar MO, Garcia DR, Oliveira MT Jr, Soeiro A, Nicolau JC, Lemos PA Neto, Rochitte CE, Ramires JA, Kalil R Filho, Porter TR. Diagnostic Ultrasound Impulses Improve Microvascular Flow in Patients With STEMI Receiving Intravenous Microbubbles. J Am Coll Cardiol. 2016 May 31;67(21):2506-15. doi: 10.1016/j.jacc.2016.03.542. PMID 27230046

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Patients With High Risk STEMI
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spontaneous Reperfusion
Description: Spontaneous reperfusion as assessed by a pre PCI ECG complete ST-segment resolution (>50%) (immediately prior to angiogram)
Time Frame: Day 1
Population: for patients did not have a pre PCI ECG
Measure: Number; unit: participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 11
participants | 2

2. Primary Outcome: Number of Participants With Spontaneous Reperfusion
Description: Spontaneous reperfusion as assessed by a pre PCI TIMI 2-3 flow on diagnostic angiogram (immediately prior to angiogram)
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
participants | 7

3. Secondary Outcome: Number of Participants With Complete (>50%) ST-segment Resolution at 30 Minutes Post PCI
Description: Complete ST-segment resolution as assessed by the worst lead on electrocardiogram (ECG core lab)
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
participants | 14

4. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) by Echocardiography (ECHO) (Simpson Method)
Description: assessed on day 1 (pre and post reperfusion), day 3±2 (discharge) and day 90±2 days after infarction
Time Frame: Day 1, Day 3±2, 3 month Follow Up
Population: EF
Measure: Mean (Standard Deviation); unit: % ejection fraction
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
% ejection fraction
  EF at 3 months | 54.9 (10.6)
  EF Day 3+/-2 | 54.6 (9.9)
  EF Day 1 post PCI | 54.5 (12.2)
  EF Day 1 pre PCI: number analyzed (Participants) | 14
  EF Day 1 pre PCI | 52.3 (10.8)
  EF Day 1 admission | 51.5 (11.6)

5. Secondary Outcome: Wall Motion Score Index (WMSI) by ECHO
Description: Mean Regional Wall Motion Score Index assessed on day 1 (pre and post reperfusion), day 3±2 (discharge) and 90±2 days after infarction. The wall motion score is determined by visual assessment of the regional wall LV wall motion in the three apical echocardiographic views. The wall motion score of LV segments is dimensionless: normal 1, hypokinetic 2, akinetic 3, dyskinetic 4. The wall motion score index is the sum of all segmental scores divided by the number of segments analyzed (scale 1-4). A wall motion score index of 1 is normal. The worse the wall motion score index the worse is the outcome.
Time Frame: Day 1, Day 3±2 , 3 month Follow Up
Population: Wall Motion Score Index (WMSI)
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
dimensionless
  WMSI 3 months: number analyzed (Participants) | 14
  WMSI 3 months | 1.4 (0.4)
  WMSI Day 3+/-2 | 1.5 (0.3)
  WMSI Day 1 post PCI | 1.6 (0.3)
  WMSI Day 1 pre PCI | 1.8 (0.3)
  WMSI Day 1 admission | 1.8 (0.3)

6. Secondary Outcome: Microvascular Perfusion Score Index (MPSI) by ECHO
Description: Mean microvascular perfusion score index (MPSI) assessed on day 1 (pre and post reperfusion), day 3±2 (discharge) and 90±2 days after infarction The microvascular perfusion score is determined by visual assessment of the LV segments in the three apical echocardiographic views. The microvascular perfusion score of LV segments is dimensionless: normal 1, mildly reduced perfusion 2, no perfusion displayed 3. The microvascular perfusion score index score index is the sum of all segmental scores divided by the number of segments analyzed (scale 1 -3). A microvascular perfusion score index of 1 is normal. The worse the microvascular perfusion score index the worse is the outcome.
Time Frame: Day 1, Day 3±2, 3 month Follow Up
Population: Microvascular Perfusion Score Index (MPSI)
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
dimensionless
  MPSI 3 months: number analyzed (Participants) | 14
  MPSI 3 months | 1.2 (0.2)
  MPSI Day 3+/-2 | 1.3 (0.3)
  MPSI Day 1 post PCI | 1.4 (0.3)
  MPSI Day 1 pre PCI | 1.6 (0.2)
  MPSI Day 1 admission | 1.7 (0.3)

7. Other Pre Specified Outcome: Number of Participants With Allergic Reaction to Definity®
Description: Number of participants who recorded any allergic reaction to Definity
Time Frame: Day 1, Day 3±2, 3 month Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
Participants | 0

8. Other Pre Specified Outcome: Number of Participants With Vasospasm in Culprit Coronary Artery
Description: Number of participants who recorded any vasospasm due to high impulse ultrasound
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
Participants | 0

9. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Number of participants who recorded any adverse events that as per protocol are not related to acute myocardial infarction
Time Frame: Day 1, Day 3±2, 3 month Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients With High Risk STEMI
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Adult Patients With High Risk STEMI
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patients With High Risk STEMI (N=15)
Ventricular Fibrillation Arrest during angiography (Cardiac disorders) | 1 (1) — Defibrillation with prompt recurrence of sinus rhythm
LV thrombus displayed at discharge echocardiogram (Cardiac disorders) | 1 (1) — Patient was admitted to initiate Warfarin treatment and intravenous heparin until therapeutic coagulation
Congestive heart failure due to severe mitral regurgitation (Cardiac disorders) | 1 (1) — Medical treatment for congestive heart failure and mitral valve replacement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patients With High Risk STEMI (N=15)
congestive heart failure (Cardiac disorders) | 2 (3) — shortness of breath, congestive was treated with furosemide and the patient improved
post myocardial infarct pericarditis (Cardiac disorders) | 1 (1)
shingles (Skin and subcutaneous tissue disorders) | 1 (1)
nausea and vomiting after morphine injection (Gastrointestinal disorders) | 1 (1)
Diplopia after angiography (Nervous system disorders) | 1 (1) — improved and patient referred to neurology
small loculated pericardial effusion (Cardiac disorders) | 1 (1)
exertional breathlessness (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03092089/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03092089/ICF_001.pdf